CLINICAL TRIAL: NCT00373945
Title: A Retrospective Case-Control Study to Estimate the Sensitivity and Specificity of a Pharmacogenetic Marker (HLA-B*5701) in Subjects With and Without Hypersensitivity to Abacavir.
Brief Title: HLA-B*5701 And Hypersensitivity To Abacavir
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: ABC107442; SHAPE
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: HIV Infection
Keywords: HLA-B*5701; pharmacogenetic marker; hypersensitivity to abacavir,; retrospective analysis
MeSH Terms: conditions — HIV Infections | interventions — Observation

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Drug: Observational Study

SUMMARY:
This retrospective case-control study is being conducted to estimate the sensitivity of the pharmacogenetic marker, HLA-B*5701 for hypersensitivity to abacavir (ABC HSR). The specificity of the marker, and its association with ABC HSR, as measured by odds ratios and 95% confidence intervals, will be evaluated as secondary endpoints. Cases will be defined in two ways - subjects who have clinically-suspected ABC HSR and a positive abacavir skin patch test reaction (CS-SPTPos) and subjects with clinically-suspected ABC HSR (CS-HSR), regardless of the results of skin patch testing. The study will include 40 CS-SPTPos Black cases matched with up to 200 abacavir-tolerant controls. In parallel, 40 CS-SPTPos White cases will be matched with up to 200 White controls. Some of the secondary analyses will use cases defined by clinical criteria alone (CS-HSR). Black and White subjects will be analyzed separately because of the differences in ABC HSR rates and in the carriage frequency of HLA-B*5701.

ELIGIBILITY:
Inclusion criteria:

* Subjects with HIV-1 infection with clinically-suspected hypersensitivity to abacavir.
* Subjects must provide consent for skin patch testing and pharmacogenetic evaluation.

Exclusion criteria:

* Women found to be pregnant at baseline.
* Subjects with HIV-1 infection who have tolerated abacavir for at least 12 weeks without experiencing hypersensitivity to the drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2006-08; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (44):
- United States (44):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Balitmore, Maryland
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Catskill, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin